CLINICAL TRIAL: NCT02436512
Title: A Phase 3 Open-label Multi-Center, Two-Part Single-arm Study to Evaluate the Acute Vasodilation Response of Inhaled Nitric Oxide as a Predictor of Successful Wean From Parental Prostacyclins in Subjects With Pulmonary Arterial Hypertension
Brief Title: Study to Assess Acute Vasodilation Response of Inhaled Nitric Oxide
Acronym: EAGLE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability meet enrollment in study population.
Sponsor: Geno LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P-2014-001
Record Dates: First submitted 2015-04-13; First posted 2015-05-06 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inhaled Nitric Oxide (Experimental): Active Comparator: Nitric Oxide
  Interventions: Drug: Inhaled Nitric Oxide

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — The investigational product is inhaled nitric oxide delivered via nasal cannula or venturi mask with the GeNOsylTM Delivery System or GeNOsylTM Acute DS, during RHC as follows:
  * (Dose 1): 5 ppm inhaled nitric oxide for 15 minutes
  * (Dose 2): 40 ppm inhaled nitric oxide for 15 minutes
  Other Names: GeNOsyl(R) Delivery System; GeNOsyl(R) Acute DS

SUMMARY:
The EAGLE study is a Phase 3, open-label, multi-center, two-part, single-arm study of GeNOsyl(R) delivery system(s) to evaluate if inhaled nitric oxide-induced vasodilation predicts successful wean from parenteral prostacyclin (PGI) in subjects with World Health Organization (WHO) Group 1 pulmonary arterial hypertension (PAH) undergoing a medically necessary right heart catheterization (RHC). All subjects enrolled in the study will undergo an attempt to wean from parenteral PGI per standard of care.

DETAILED DESCRIPTION:
This study will be divided into 2 parts: a Pilot Phase followed by Pivotal Phase.

* The Pilot Phase will enroll up to 20 subjects. The information derived from the Pilot Phase will evaluate safety, and assess the vasoreactivity test response rate.
* Approximately 150 subjects will be enrolled in the Pivotal Phase of the study, to gather further data on weaned successes from parenteral PGI. The Investigator and study staff involved with the wean and patient management will be blinded in this phase of the study to the vasoreactivity results.

ELIGIBILITY:
Inclusion Criteria:

* The subject or subject's legally authorized representative signs and dates an Institutional Review Board (IRB) approved informed consent form prior to the initiation of any study-related activities.
* The subject has been diagnosed with PAH (WHO Group 1) and is WHO Functional Class I or II at Screening.
* The subject has documented continuous PGI use for ≥ 1 year from Screening, without a significant interruption (i.e., ≤ 2 day interruption) and without a failed complete wean attempt.
* The subject is a candidate for weaning off parenteral PGI therapy (per Investigator judgment and standard of care).

Exclusion Criteria

* The subject has a hypersensitivity or allergy to ingredients of inhaled nitric oxide or other clinically significant allergies (clinical significance per Investigator judgment).
* The subject has a PCWP or left ventricular end diastolic pressure (LVEDP) ≥15 mmHg at Baseline.
* The subject has participated in an investigational product or device study within the 30 days prior to Screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Wean Success vs Wean Failure | Visit 4 - Day 84
  To evaluate the number of subjects that achieve Wean Success that are Vasoreactivity Response (VR) positive (+) versus VR negative (-)and the number of subjects that are Wean Failures that are VR(+) versus VR(-).
  Wean-Success:
  * No parenteral PGI therapy at 3 months post-wean completion; and
  * Clinical stability, where clinical stability is defined as:
    * A decrease in 6MWT distance less than 10% from pre-wean; and
    * NT-proBNP increase <15% from pre-wean; and
    * WHO Functional Class <III
  Wean-Failure:
  * Subjects that wean successfully but do not meet all clinical stability components of the Wean-Success definition above; or
  * Failure to wean within the 3 month Transition Period; or
  * Re-initiation of parental PGI during the 3 month post-wean or subject does not meet the definition of clinical stability at 3 month post-wean; or
  * Death or hospitalization due to progression of disease; or
  * Atrial septostomy; or
  * Heart and/or lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Cassie Newell, MAOM, Study Director — Geno LLC
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - Allegheny General Hospital, Pittsburgh, Pennsylvania